CLINICAL TRIAL: NCT04310826
Title: Feasibility of Dietary Magnesium Replacement for Prevention of Hypomagnesemia in Ovarian Cancer Patients Receiving Carboplatin Chemotherapy
Brief Title: Dietary Magnesium in Preventing Low Blood Magnesium Levels in Patients With Ovarian Cancer Receiving Carboplatin Chemotherapy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2018-1172; NCI-2019-02450 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-1172 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-03-13; First posted 2020-03-17 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Ovarian Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prevention (dietary intervention) (Experimental): Patients receive a dietary magnesium intervention consisting of a food reference list and phone calls or video interviews from a registered dietitian, integrative medicine physician, or a mid-level provider over 10-20 minutes once a week for up to the 6th cycle of chemotherapy (average 15 weeks).
  Interventions: Dietary Supplement: Dietary Intervention; Other: Media Intervention; Behavioral: Telephone-Based Intervention

INTERVENTIONS:
Dietary Supplement: Dietary Intervention — Receive dietary magnesium intervention
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions
Other: Media Intervention — Undergo video interviews
Behavioral: Telephone-Based Intervention — Receive phone calls

SUMMARY:
This trial studies how well a diet high in magnesium works in preventing low blood magnesium levels (hypomagnesemia) in patients with ovarian cancer receiving carboplatin chemotherapy. Hypomagnesemia is a common side effect of carboplatin-containing chemotherapy. A magnesium rich diet may increase the levels of magnesium in the blood and help prevent hypomagnesemia resulting from carboplatin chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate intervention feasibility.

SECONDARY OBJECTIVE:

I. Evaluate occurrence of hypomagnesemia and the need for a pharmacy regimen including oral and intravenous magnesium dosage.

EXPLORATORY OBJECTIVE:

I. Explore changes in other electrolytes, weight, and occurrence of chemotherapy delay or discontinuation and hospitalization which can be related to dietary intervention and program completion.

OUTLINE:

Patients receive a dietary magnesium intervention consisting of a food reference list and phone calls or video interviews from a registered dietitian, integrative medicine physician, or a mid-level provider over 10-20 minutes once a week for up to the 6th cycle of chemotherapy (average 15 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Patients with previously untreated ovarian cancer.
* Receiving carboplatin-containing chemotherapy of at least 6 consecutive cycles.
* Able to tolerate an oral diet.

Exclusion Criteria:

* Prior platinum-based chemotherapy.
* Serum creatinine level > 1.4 mg/dL prior to treatment.
* Artificial nutrition (e.g. Ensure or Boost) accounts for > 50% of total calorie intake.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Patient retention rate | Up to 2 years
  Assessed by percentage of patients completing the dietary intervention. If a patient participated 60% or more of the weekly follow up by the end of the 6th cycle of treatment, she is considered retained. Descriptive statistics (e.g., frequencies, proportions, means, standard deviations [SDs], and ranges), along with 95% confidence intervals (CIs) for the means, will be computed.
Dietary adherence rate | Up to 2 years
  Ratio of actual dietary magnesium intake versus the desired 400 mg. Descriptive statistics (e.g., frequencies, proportions, means, SDs, and ranges), along with 95% CIs for the means, will be computed.

SECONDARY OUTCOMES:
Occurrence of hypomagnesemia | Up to 2 years
  Descriptive statistics (e.g., frequencies, proportions, means, SDs, and ranges), along with 95% CIs for the means, will be computed.
Need for a pharmacy intervention including oral and intravenous magnesium dosage | Up to 2 years
  Descriptive statistics (e.g., frequencies, proportions, means, SDs, and ranges), along with 95% CIs for the means, will be computed.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Cohen, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2022-03-28): https://cdn.clinicaltrials.gov/large-docs/26/NCT04310826/ICF_000.pdf